CLINICAL TRIAL: NCT02973178
Title: Scanadu Urine Device Validation Study Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scanadu, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FO-004
Record Dates: First submitted 2016-11-15; First posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Urinary Tract Infections; Proteinuria; Ketone Urine; Hematuria; Glucose Intolerance
MeSH Terms: conditions — Urinary Tract Infections; Proteinuria; Ketosis; Hematuria; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usability (Other): Evaluate and validate the user-interface of the Scanadu Urine Device by the intended users for human factors and user interface of the Scanadu Urine Device.
  Interventions: Device: Scanadu Urine Device
- Method Comparison (Active Comparator): Evaluate and validate the clinical performance of the Scanadu Urine Device in the hands of intended users as compared to:
  * The visual read of chemical test strips performed by lab technicians utilizing the Siemens Multistix® 10SG technology (K905396),
  * Scanadu Urine Device tests performed by lab technicians.
  Interventions: Device: Scanadu Urine Device
- Reproducibility (Other): Evaluate the reproducibility in the hands of the lay-users after repeated testing of samples with known test levels.
  Interventions: Device: Scanadu Urine Device

INTERVENTIONS:
Device: Scanadu Urine Device — Device to allow lay user to perform urinalysis test at home.

SUMMARY:
This study will test Scanadu Urine Device for clinical performance and usability.

DETAILED DESCRIPTION:
The objectives of this study are to:

* Evaluate and validate the clinical performance of the Scanadu Urine Device in the hands of intended users as compared to: the visual read of chemical test strips performed by lab technicians utilizing the Siemens Multistix® 10SG technology (K905396).
* Evaluate and validate the user-interface of the Scanadu Urine Device by the intended users for human factors and user interface of the Scanadu Urine Device.
* Evaluate the reproducibility in the hands of the lay-users after repeated testing of samples with known test levels

ELIGIBILITY:
Inclusion Criteria:

* Female and male
* 18 years old or older
* Pregnant or not pregnant
* Must have experience using an Apple iPhone
* Have no visual impairments
* Able to hold Smart Phone horizontally in raised dominant hand
* Must be able to read and understand English
* Must provide Informed Consent

Exclusion Criteria:

* Has a known history of a visual impairment that may affect reading and navigating the Scanadu Urine app
* Unable to void and collect urine specimen for testing
* Unable to hold phone steady (horizontally) or has history of tremors or conditions such as Parkinson's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Usability: % successful scans in three tests conducted by lay users in following the app on the iPhone and obtain user experience on questionnaire | Single visit in one day
  Evaluate and validate the user-interface of the Scanadu Urine Device by the intended users for human factors and user interface of the Scanadu Urine Device.
Method Comparison: Conduct two tests by following iPhone app (self and patient samples), results in concordance with professional testers; achieve accuracy in different concentrations of six urine analytes each using approximately 20 samples per level. | Single visit in one day
  Evaluate and validate the clinical performance of the Scanadu Urine Device in the hands of intended users as compared to: the visual read of chemical test strips performed by lab technicians utilizing the Siemens Multistix® 10SG technology (K905396).
Reproducibility: Lay user's ability to repeat a urine test nine times by following iPhone app and obtain nine results that are in concordance. | Single visit in one day
  Evaluate the reproducibility in the hands of the lay-users after repeated testing of samples with known test levels

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - West Coast Research, LLC, Mountain View, California
  - West Coast Research, LLC, San Leandro, California

IPD SHARING:
Plan to Share IPD: No